CLINICAL TRIAL: NCT01491620
Title: A Single-Center Prospective, Open-Label Study of the Excel V 532 nm KTP Laser for the Treatment of Poikiloderma of Civatte
Brief Title: Study of the 532 nm KTP Laser for the Treatment of Poikiloderma of Civatte
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cutera Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C-11-XPC01
Record Dates: First submitted 2011-12-05; First posted 2011-12-14 (Estimated); Results first posted 2022-10-28 (Actual); Last update posted 2022-10-28 (Actual); Status verified 2022-10

CONDITIONS: Poikiloderma of Civatte; Dyschromia; Pigmentation Disorders; Telangiectasia; Photosensitivity Disorders
Keywords: poikiloderma of Civatte; red dyschromia; brown dyschromia; sun damage; neck; chest; dyschromia; pigmentation disorders; erythema; photosensitivity disorders; sun exposure; telangiectasia; hyperpigmentation; hypopigmentation
MeSH Terms: conditions — Pigmentation Disorders; Telangiectasis; Photosensitivity Disorders; Erythema; Hyperpigmentation; Hypopigmentation | interventions — Lasers, Solid-State

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- 532 nm KTP laser treatment (Experimental)
  Interventions: Device: 532 nm KTP laser

INTERVENTIONS:
Device: 532 nm KTP laser — Laser treatment sessions on the neck and/or chest
  Other Names: Excel V

SUMMARY:
This study will evaluate the safety and efficacy of the Excel V 532 nm KTP laser for the treatment of dyschromia of the neck and/or chest (poikiloderma of Civatte).

ELIGIBILITY:
Inclusion Criteria:

* Fitzpatrick Skin Type I - III
* Clinical diagnosis of poikiloderma of Civatte affecting the neck and/or chest
* Willing to refrain from using topical corticosteroids, retinoids and bleaching agents on the treated area
* Agree not to undergo any other procedure for the treatment of poikiloderma of Civatte during the study
* Willing and able to read, understand and sign the Informed Consent Form
* Willing and able to adhere to the treatment and follow-up schedule and post-treatment care instructions

Exclusion Criteria:

* Any laser treatment on neck and/or chest within 12 months
* Any topical treatment on neck and/or chest within 6 months
* Pregnant and/or breastfeeding
* Infection, dermatitis or a rash in the treatment area
* Suffering from significant concurrent illness, such as Diabetes Mellitus or pertinent neurological disorders
* History of seizure disorders due to light, fibromyalgia, connective tissue disease, vitiligo, psoriasis, pigmentary disorders, keloid scarring, hypertrophic scarring or abnormal wound healing
* History of immunosuppression/immune deficiency disorders or currently using immunosuppressive medications
* Having a known anticoagulative condition or taking anticoagulation medications
* History of diseases stimulated by heat, unless treatment is conducted following a prophylactic regimen
* Having undergone any surgery in the treatment area within 6 months of treatment (or more if skin has not healed completely)
* History of radiation to the head, neck and/or upper chest
* Undergoing systemic chemotherapy for the treatment of cancer
* Systemic use of isotretinoin (Accutane®) within 6 months
* Any use of gold therapy
* Excessively tanned in areas to be treated or unable/unlikely to refrain from tanning during the study
* Current smoker or history of smoking within 12 months of study
* Participation in a study of another device or drug within 6 months
* As per the Investigator's discretion, any physical or mental condition which might make it unsafe for the subject to participate in study

Ages: 35 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2011-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Zel Skin and Laser Specialists, Edina, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- 532 nm KTP Laser Treatment: 532 nm KTP laser: Laser treatment sessions to neck and/or chest.
Period: Overall Study
Arm/Group | 532 nm KTP Laser Treatment
Started | 24
Completed | 24
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- 532 nm KTP Laser Treatment: 532 nm KTP laser: Two laser treatment sessions to neck and/or chest. 6 weeks apart.
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 24
Age, Continuous [Mean (Full Range); unit: years] | 52.5 [40 to 64]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 24
  Male | 0

OUTCOME MEASURES:

1. Primary Outcome: Severity Assessment Score
Description: Change in Physician's Severity Assessment score based on blinded assessment of subject photographs by a panel of independent dermatologists.
  Blinded Physician's Severity Assessment (min=1;max=4); Higher scores mean worse values
Time Frame: 24 weeks
Population: Only 5 subjects were treated and then assessed at 24 weeks in their upper chest area
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 17
score on a scale
  Neck | -0.06 (0.66)
  Upper Chest: number analyzed (Participants) | 5
  Upper Chest | 0.2 (0.45)

2. Primary Outcome: Physician's Global Assessment (Blinded)
Description: Before and after subject photographs were presented to a panel of independent dermatologists. The panel was blinded to treatment parameters and the photograph time points. Each dermatologist was asked to select the baseline photograph and then rate improvement in Poikiloderma of Civatte in the post-treatment photograph using a 5-point improvement scale.
  Physician's Global Assessment (min= -1; max=4) Higher scores mean better outcome
Time Frame: 24 weeks
Population: Only 5 subjects were treated and then assessed at 24 weeks in their upper chest area
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | 532 nm KTP Laser Treatment
Number analyzed (Participants) | 17
score on a scale
  Neck Area | .06 (.97)
  Upper Chest Area: number analyzed (Participants) | 5
  Upper Chest Area | 1 (.71)

ADVERSE EVENTS:
Groups:
- 532 nm KTP Laser Treatment: 532 nm KTP laser: Laser treatment sessions to neck or chest
Arm/Group | 532 nm KTP Laser Treatment
All-Cause Mortality (participants affected / at risk) | 0/24
Serious Adverse Events (participants affected / at risk) | 0/24
Other Adverse Events (participants affected / at risk) | 24/24
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | 532 nm KTP Laser Treatment (N=24)
Erythema (Skin and subcutaneous tissue disorders) | 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No